CLINICAL TRIAL: NCT02162303
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Colchicine on Vascular Inflammation as Assessed With Position Emission Tomography (PET) Imaging in Patients With Atherosclerotic Vascular Disease (COLPET)
Brief Title: Colchicine in Vascular Inflammation Assessed With PET Imaging
Acronym: COLPET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MHIPS-002
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Atherosclerotic Vascular Disease
Keywords: Atherosclerosis; Vascular; Cardiovascular; Coronary artery disease; Imaging; PET; Scan; anti-inflammatory
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Colchicine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine 0.6 mg tablets,once daily, for 6 months
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Sugar,given once daily, over 6 months.To mimic active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 0.6 mg a day of active treatment or placebo for 24 weeks
  Other Names: Colchicum autumnale
  Arms: Colchicine
Drug: Placebo — Sugar,given once daily, over 6 months.To mimic active treatment
  Other Names: Sugar
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the effects of colchicine on vascular inflammation measured by (FDG)-PET imaging in patients with atherosclerotic vascular disease. This effect will also be measured by soluble plasma biomarkers. Finally, an optional pharmacogenomic investigation will be performed to identify genetic biomarkers of patient response.

DETAILED DESCRIPTION:
This is an interventional trial targetting patients 18 years old or older with a carotid artery or an ascending aorta to background ration (TBR) of ≥1.6 as determined by 18 fluorodeoxyglucose (18F-FDG) uptake measured by positron emission tomography (PET) as evidence of atherosclerotic plaque inflammation.

Following randomization,patients will be followed over a period of 6 months (24 weeks), through 2 phone contacts at 6 and 20 weeks and 2 on-site visits at 12 and 24 weeks.

Each on-site visits will include blood draws to monitor routine chemistry and hematology,as well as biomarkers and lipid profiles.

Each phone contacts will include monitoring of patient's general health and well-being.

PET imaging will be performed at baseline and at the 24-weeks visit.

Safety in this study will be assessed by clinical laboratory parameters, physical examinations, ECGs, vital signs, and the frequency and intensity of clinical adverse events (AEs).

The Montreal Health Innovations Coordinating Center (MHICC) will be responsible for processing and quality control of the data. Project management will be carried out as described in the MHICC standard operating procedures (SOPs) for clinical studies. The handling of data, including data quality control, will comply with all applicable regulatory guidelines, MHICC SOPs and the study Data Management Plan. As such, a MHICC medical monitor will be appointed to the trial as the serious adverse event reporting contact (24/7).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients providing informed consent
* Patient must have evidence of coronary artery disease (CAD) as evidenced by at least one of the following:
* Angiographic evidence of at least 50% stenosis in one coronary artery (except for left main coronary artery stenosis, in which 30% is acceptable)
* History of prior percutaneous coronary intervention (PCI)
* History of prior acute coronary syndrome (ACS) event (ST elevation myocardial infarction (STEMI), non-STEMI or unstable angina)
* Patient has a carotid or ascending aorta atherosclerotic plaque inflammation TBR of 1.6 or more as determined by 18F-FDG uptake measured by PET scanning
* Patient must be on a stable dose for at least 8 weeks before baseline if taking medications used to control angina, hypertension, serum lipids (including statins) or any medication that can have an effect on inflammation
* Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practices a birth control method throughout the study and for 30 days after study completion
* Patient is judged to be in good general health as determined by the principal investigator
* Patient must be able and willing to comply with the requirements of this study protocol

Exclusion Criteria:

Poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, congestive heart failure, a left ventricular ejection fraction of less than 40%, recent stroke (within the past 3 months), chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study

* History of ACS, PCI, myocardial infarction, carotid revascularization or hospitalization for a cardiac condition within 12 weeks of baseline
* Prior coronary artery bypass graft
* Planned change in medical treatment during the study, that can have effect on inflammation, for angina, serum lipids, and other conditions
* History of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* History of listeriosis, treated or untreated tuberculosis, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infective agent within 30 days or oral anti-infective agent within 14 days prior to baseline
* Hepatitis B or hepatitis C viral infection
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis) or patient with chronic diarrhea
* Pre-existent progressive neuromuscular disease or patient with creatine phosphokinase (CPK) level > 3 times the upper limit of normal at baseline
* Current use or plans to use anti-retroviral therapy at any time during the study, or with active chronic disease often treated with a protease inhibitor, including AIDS
* Diagnosed with immune deficiency or as immunocompromised
* Any of the following: hemoglobin < 120g/L, white blood cell count < 3.0 X 109/L, platelet count <130 X 109/L, Alanine aminotransferase (ALT) > 3 times the upper limit of normal, Aspartate aminotransferase (AST) > 3 times the upper normal limit, total bilirubin > 2 times the upper normal limit, creatinine > 150 umol/L, creatinine clearance < 30 mL/min, or history of cirrhosis or severe hepatic disease
* Pregnant or breast-feeding or considering becoming pregnant during the study or for 6 months after the last dose of study medication
* History of clinically significant drug or alcohol abuse in the last year
* Previous bilateral carotid surgery
* Other indications for colchicine use (mainly chronic indications represented by Familial Mediterranean Fever or gout)
* History of an allergic reaction or significant sensitivity to constituents of study drug
* Use of an investigational chemical agent less than 50 days or 5 half-lives prior to baseline (whichever is longer)
* Judged by the investigator to be an unsuitable candidate for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in the average of maximum target-to-background (TBR) values (Mean MAX TBR) of the ascending aorta | baseline and 6 months

SECONDARY OUTCOMES:
Change in the Mean Maximum Target-to-background (Mean MAX TBR) of carotid arteries | baseline and 6 months
Change in the average of the mean TBR values (Mean MEAN TBR) | baseline and 6 months
Change in the Most Diseased Segment TBR values (MDS TBR) in the carotid arteries and ascending aorta | baseline and 6 months
  MDS TBR is defined as the 1.5 cm segment that demonstrates the highest PET/CT activity at baseline and is calculated as the Mean Max TBR values derived from approximately 5 contiguous axial segments.
Change in soluble biomarkers of inflammation | baseline and 6 months
  Soluble biomarkers of inflammation include high sensitivity C-Reactive Protein (hs-CRP). As well, frozen samples (whole blood, plasma and leucocytes for RNA analyses) will be kept for future use for evaluation of biomarkers related to cardiovascular disease and responses to the treatment mostly regarding: lipid, inflammation and oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided